CLINICAL TRIAL: NCT06905652
Title: Comparative Acute Effects of R-MDMA and S-MDMA in Healthy Participants
Acronym: R-S-
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2024-01835
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: double-blind, placebo-controlled, 3-period cross-over design with two treatment conditions and placebo: 1. R-MDMA (300mg), 2. S-MDMA (100mg), 3. Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 300mg R-MDMA (Experimental): R-MDMA (300mg)
  Interventions: Drug: R-3,4-methylenedioxymethamphetamine
- 100mg S-MDMA (Experimental): S-MDMA (100mg)
  Interventions: Drug: S-3,4-methylenedioxymethamphetamine
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: R-3,4-methylenedioxymethamphetamine — A dose of 300mg enantiomeric R-MDMA will be administered.
  Other Names: R-MDMA
  Arms: 300mg R-MDMA
Drug: S-3,4-methylenedioxymethamphetamine — A dose of 100mg enantiomeric S-MDMA will be administered.
  Other Names: S-MDMA
  Arms: 100mg S-MDMA
Other: Placebo — Placebo (Mannitol)
  Arms: Placebo

SUMMARY:
Racemic ±3,4-methylenedioxymethamphetamine (MDMA) is a psychoactive substance and prototypical empathogen acutely inducing feelings of heightened mood, empathy, trust and closeness to others. These acute subjective effects of MDMA may be helpful to assist psychotherapy and MDMA has been investigated in phase 3 trials as a possible treatment in post-traumatic stress disorder.

DETAILED DESCRIPTION:
MDMA is a racemic substance containing equal amounts of the enantiomers S(+)- and R(-)-MDMA. Preclinical research indicates that S-MDMA mainly releases dopamine (DA), norepinephrine (NE), serotonin (5-HT), and oxytocin while R-MDMA may act more directly on 5-HT2A receptors and release prolactin (PRL). Animal studies also indicate that the two enantiomers act synergistically to produce the subjective effects of MDMA and that S-MDMA is mainly responsible for psychostimulation while R-MDMA may have fewer adverse effects and have greater prosocial effects. A human study conducted between 10/2022 and 01/2024 by our team compared the effects of R-MDMA, S-MDMA, and racemic MDMA revealing that both enantiomers have generally similar effects. However, the study did not administer equivalent doses of R- and S-MDMA. In the present study a single dose of R-MDMA and a single dose of S-MDMA, now adjusted and presumed to be equivalent, will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. Good understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Willing not to operate heavy machinery within 48 h after administration of a study substance (including driving a car)
7. Willing to use effective birth-control throughout study participation.
8. Body mass index 18 - 34.9 kg/m2

Exclusion Criteria:

1. Relevant chronic or acute medical condition
2. Current or previous major psychiatric disorder (e.g. bipolar disorder, schizophrenia), current depression or anxiety disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Illicit substance use (not including cannabis) more than 20 times or any time within the previous month.
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medications that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day).
10. Excessive consumption of alcoholic beverages (>15 drinks/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Subjective effects | through study completion, an average of 18 months.
  Any drug effect on the Visual Analog Scales (VAS) assessing the intensity and duration of the subjective effect on a scale from 0 - 100 percent with higher scores representing more intense effects 14 times each study day.

SECONDARY OUTCOMES:
Autonomic effects I | Through study completion, an average of 18 months.
  Blood pressure (systolic and diastolic) will be measured with an automatic oscillometric device 14 times each study day.
Autonomic effects II | Through study completion, an average of 18 months.
  Heart rate will be measured with an automatic oscillometric device. Assessed 14 times on each study day.
Autonomic effects III | through study completion, an average of 18 months.
  Body temperature will be measured with an ear thermometer. Assessed 14 times each study day.
Plasma levels of oxytocin | Through study completion, an average of 18 months.
  Assessed 3 times on each study day
Plasma levels of cortisol | Through study completion, an average of 18 months.
  Assessed 3 times on each study day
Plasma levels of prolactin | Through study completion, an average of 18 months.
  Assessed 3 times on each study day
Plasma levels of R-MDMA | Through study completion, an average of 18 months.
  Assessed 13 times on each study day
Plasma levels of S-MDMA | Through study completion, an average of 18 months.
  Assessed 13 times on each study day
Additional subjective effects I | Through study completion, an average of 18 months.
  Visual Analog Scales (VAS) assessing the intensity and duration of subjective effects on a scale from 0 - 100 percent with higher scores representing more intense effects. Assessed 14 times on each study day
Additional subjective effects II | Through study completion, an average of 18 months.
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely" assessed 4 times on each study day
Additional subjective effects III | Through study completion, an average of 18 months.
  This world connectogen scale (TWCS) assessing the connectogenic properties of MDMA as a strong sense of connection with the here-and-now, the body, the world and spiritual principles. Assessed once each study day
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Freiburger Personality Inventory (FPI-R) | Baseline
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücken Personality Questionnaire (SPF) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Saarbrücker Persönlichkeitsfragebogen (SPF) defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
HEXACO personality inventory | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Defense Style Questionnaire (DSQ-40) | Baseline
  Personality traits are known to affect subjective responses to psychoactive substances and are assessed for explorative future analysis of pooled data. The Defense Style Questionnaire (DSQ-40) can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".
Acute adverse effects | Through study completion, an average of 18 months.
  Assessed twice on each study day with the list of complaints (LC)
Subacute adverse effects I | Through study completion, an average of 18 months.
  The List of complains is a list of 50 symptoms assessed on a 4-point Likert scale ranging from "not at all" to "extremely". Assessed twice (24 and 72h) after each study day.
Subacute adverse effects II | Through study completion, an average of 18 months.
  The Beck Depressionindex questionnaire (BDI) is assessed once after each study day (72h) with low values indicating normal mood and high values indicating severe depression.
Dose equivalence I | Through study completion, an average of 18 months.
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects with higher scores representing more intense effects. Assessed once on each study day
Dose equivalence II | Through study completion, an average of 18 months.
  The State of Consciousness (SCQ) Questionaire assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely") once on each study day
Life satisfaction and well-being I | Through study completion, an average of 18 months.
  The Scale of positive and negative experience (SPANE) assesses 12 items of subject well-being on a 5-point-scale ranging from "very rarely" to "very often or always". Assessed once each study day and 72 h after administration.
Life satisfaction and well-being II | Through study completion, an average of 18 months.
  The "positive attitude towards life" is an 8-item subscale of the Berner Subjective Well-Being Quetsionaire for adults (BFW/E) using a six-point rating scale from "strongly disagree" (1) to "strongly agree" (6) to rate the attitude towards life. Assessed once each study day.
Life satisfaction and well-being III | Through study completion, an average of 18 months.
  The Global Life Satisfaction (GLS) assesses the overall satisfaction on a 11 point scale with 0 meaning "not at all satisfied" and 10 meaning "completely satisfied". Assessed once each study day as well as 72 h after each drug adminstration.
Life satisfaction and well-being IV | Baseline/End of Study Visit
  The Appreciation Scale (AS) includes 57 items to measure eight aspects of appreciation. Subjects are asked to rate themselves on a scale from 1 to 7 in terms of either attitude intensity ('strongly disagree' to 'strongly agree') or frequency ('never' to 'more than once a day'). Assessed at screening and end of study visit.
Empathogenic effects I | Through study completion, an average of 18 months.
  Multifaceted Empathy Test (MET), effects on empathy in computer tests, assessed one time during each study session.
Empathogenic effects II | Through study completion, an average of 18 months.
  Facial expression recognition test (FERT), effects on empathy in computer tests, assessed one time during each study session.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland